CLINICAL TRIAL: NCT01218789
Title: Open-Label Safety Study of a 1-Year 20 mg Dose Regimen of Tasimelteon for Treatment of Non-24-Hour-Sleep-Wake Disorder (N24HSWD) in Blind Individuals With No Light Perception
Brief Title: Safety Study of Tasimelteon for Treatment of Non-24-Hour-Sleep-Wake Disorder in Blind Individuals With No Light Perception
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VEC-162-3202
Record Dates: First submitted 2010-09-28; First posted 2010-10-11 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Non 24 Hour Sleep Wake Disorder
Keywords: Blindness; Eye Diseases; Nap Disorders; Circadian Rhythm Disorders; Sleep disorders; Circadian Rhythm Sleep Disorders; Dyssomnias; Nervous System Diseases
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Blindness; Eye Diseases; Chronobiology Disorders; Sleep Wake Disorders; Dyssomnias; Nervous System Diseases | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tasimelteon (Experimental): 20 mg tasimelteon capsules, PO daily for 1 year
  Interventions: Drug: tasimelteon

INTERVENTIONS:
Drug: tasimelteon — 20 mg tasimelteon capsules, PO daily for 1 year
  Other Names: VEC-162

SUMMARY:
The purpose of this study is to evaluate the safety of a one year open-label treatment of tasimelteon in male and female subjects with Non-24-Hour Sleep-Wake Disorder.

DETAILED DESCRIPTION:
Non-24-Hour Sleep-Wake Disorder (N24HSWD) occurs when individuals, primarily those without light perception, are unable to synchronize their endogenous circadian pacemaker to the 24-hour light-dark cycle, and the timing of their circadian rhythm instead reflects the intrinsic period of their endogenous circadian pacemaker. As a result, the circadian rhythm of sleep-wake propensity in these individuals moves gradually later and later each day if there circadian period is > 24 hours and earlier and earlier if < 24 hours. These individuals will be able to sleep well at night when their sleep-wake propensity rhythm is approximately aligned with the 24-hour light-dark and social cycle. However, after a short time, the endogenous sleep-wake propensity rhythm and the 24-hour light-dark cycle will move out of synchrony with each other, and they may have difficulty falling asleep until well into the night. In addition to problems sleeping at the desired time, the subjects experience daytime sleepiness and daytime napping.

This will be a multicenter, open-label study. The study has two phases: the screening phase and the evaluation phase. The screening phase is comprised of a screening visit where a patient's general health and initial eligibility will be evaluated. The evaluation phase is comprised of a baseline visit and a 52 week segment. Patients that meet all entry criteria for the study at baseline visit will enter the treatment segment where patients will be asked to take 20 mg tasimelteon daily approximately 60 minutes prior to their target bedtime for 52 weeks in an open-label fashion. An optional sub-study extension phase is available to subjects who complete the first year of treatment and consists of continued open-label treatment for up to 3 years additional.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide informed consent;
* No perception of light;
* History (within the last 3 months) of trouble sleeping at night difficulty initiating sleep or staying asleep), difficulty awakening in the morning, or daytime sleepiness as determined by answering yes to at least one question in the Sleep Complaint Questionnaire
* Willing and able to comply with study requirements and restrictions including a commitment to a fixed 9-hour sleep opportunity during the study;

Exclusion Criteria:

* Have a probable diagnosis of a current sleep disorder other than N24HSWD that is the primary cause of the sleep disturbance based on clinical investigator medical judgment;
* Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction unless currently controlled and stable;
* History (within the 12 months prior to screening) of psychiatric disorders including Major Depressive Disorder, Generalized Anxiety Disorder, Axis II Disorders, delirium or any other psychiatric disorder that in the opinion of the clinical investigator would affect participation in the study or full compliance with study procedures;
* History of intolerance and/or hypersensitivity to melatonin or melatonin agonists;
* Smoke more than 10 cigarettes/day
* Participation in a previous tasimelteon (aka VEC-162 or BMS-214778) trial;
* Use of central nervous system prescription or OTC medications, other than melatonin, that affects the sleep-wake cycle within 3 weeks or 5 half-lives (whichever was longer) of Baseline;
* Use of melatonin or melatonin agonist;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-10-28 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluations | Week 4
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 8
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 12
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 16
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 26
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 34
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 42
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.
Safety Evaluations | Week 52
  the recording of adverse events (AEs), clinical laboratory evaluations including labs, vital signs, and electrocardiograms(ECGs).
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal behavior and ideation.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGI-C) | Weeks 8, 16, 26, 34, 42, 52
  A patient rated assessment of reported nighttime sleep
Clinical Global Impression of Change (CGI-C) | Weeks 8, 16, 26, 34, 42, 52
  rate of total improvement due to drug as viewed by the clinician
Patient Global Impression of Change (PGI-C) | Weeks 8, 16, 26, 34, 42, 52
  A patient rated assessment on daytime naps

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Garches
  - Lille
  - Lyon
  - Montpellier
  - Paris
  - Rennes
  - Toulouse